CLINICAL TRIAL: NCT03706170
Title: Emotion Assessment to Study Consciousness in Awakening Patients
Acronym: EmotiCones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL18_0622; 2018-A02673-52 (Other: ID-RCB)
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Persistent Vegetative State
Keywords: Persistent Vegetative State; minimally conscious state; Emotions; Awareness; electrodermal activity; Electroencephalography
MeSH Terms: conditions — Persistent Vegetative State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vegetative State (Experimental): For patients in vegetative state (n=15), three experiments will be performed during 2 days in order to assess emotions and consciousness with physiological variables and electroencephalography.
  Interventions: Behavioral: Physiological recording in response to different types of stimuli; Behavioral: EEG recording in response to different types of stimuli
- Minimally Conscious State (Experimental): For patients in minimally conscious state (n = 15), three experiments will be performed during 2 days in order to assess emotions and consciousness with physiological variables and electroencephalography.
  Interventions: Behavioral: Physiological recording in response to different types of stimuli; Behavioral: EEG recording in response to different types of stimuli
- Acquired Brain damaged patients without DOC (Experimental): Acquired Brain damaged patients without disorder of consciousness (patients without DOC) For patients with acquired brain damage without disorder of consciousness (n=15), three experiments will be performed during 2 days in order to assess emotions and consciousness with physiological variables and electroencephalography
  Interventions: Behavioral: Physiological recording in response to different types of stimuli; Behavioral: EEG recording in response to different types of stimuli
- Healthy subjects (Experimental): For healthy subjects (n=15), three experiments will be performed during 2 days in order to assess emotions and consciousness with physiological variables and electroencephalography.
  Interventions: Behavioral: Physiological recording in response to different types of stimuli; Behavioral: EEG recording in response to different types of stimuli

INTERVENTIONS:
Behavioral: Physiological recording in response to different types of stimuli — In order to answer these questions, the study is designed to record in a single session: (i) physiological vegetative reactions (electrodermal, pupillary responses and heart rate) to emotional stimuli ; (ii) a neurophysiological marker of consciousness; and (iii) physiological parameters during a trace conditioning experiment using auditory stimuli with and without emotional valence.
Behavioral: EEG recording in response to different types of stimuli — In order to answer these questions, the study is designed to record in a single session: (i) physiological vegetative reactions (electrodermal, pupillary responses and heart rate) to emotional stimuli ; (ii) a neurophysiological marker of consciousness; and (iii) physiological parameters during a trace conditioning experiment using auditory stimuli with and without emotional valence.

SUMMARY:
After a coma, one important challenge is the detection of awareness with patients with disorders of consciousness. For some patients, the only behavioral manifestation indicative of awareness is an appropriate emotional response. Studies show that the use of a particular conditioning - with delay - appears to be an objective solution to study the conscious perception of an emotion in none-communicating people. Until now, emotions of patients suffering disorder of consciousness (DOC) have been scarcely studied. It has been proved that some awakening patients have vegetative reactions following an emotional stimulus, but the investigator can't confirm whether or not the emotional experience of the patient is conscious.

The investigator's main purpose is to study emotional reactions from patients suffering a disorder of consciousness.

The investigator hypothesize that some patients have preserved reflexes reaction to the emotional stimuli while others could demonstrate a conscious emotional experience.

In order to answer these questions, the study is designed to record in a single session: (i) physiological vegetative reactions (electrodermal, pupillary responses and heart rate) to emotional stimuli both in DOC patients and healthy controls; (ii) a neurophysiological marker of consciousness; and (iii) physiological parameters during a trace conditioning experiment using auditory stimuli with and without emotional valence. The investigator plan to include patients vegetative patients (n=15); minimally conscious patients (n=15); acquired brain injured patients without conscious disorder (n=15) and healthy participants (n=15).

ELIGIBILITY:
Inclusion Criteria:

For Patients :

* age between 18 and 80
* acquired brain lesion (brain injury, stroke, anoxia) with a delay since the insult superior to 1 month
* level of consciousness assessed with the coma recovery scale revised (CRS-R)
* patient with health insurance
* informed consent signed by the patients or his representative

For Healthy participants:

* age between 18 and 80
* participant able to understand instructions and normal hearing
* patient with health insurance
* informed consent signed

Exclusion Criteria:

For Patients :

* non controlled epilepsy
* dysautonomic crisis
* unstable medical state
* pregnancy or breath feeding for women
* Persons under guardianship, curatorship

For Healthy participants:

* neurological disorder
* pregnancy or breath feeding for women
* Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of rights or liberty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
electrodermal response | at Day 1
  skin conductance response measured with trans-cutaneus electrodes

SECONDARY OUTCOMES:
pupillary response | at Day 1
  use of eye-tracker
heart rate modification | at day 1
  use of transcutaneous electrode
Variation of the intensity of different Event Related Potentials | at Day 2
  electroencephalography (EEG) The investigator will study how the intensity of different Event Related Potentials varies with different levels of sound around the auditory threshold: this will be assessed specifically for early cortical components of the auditory response such as the N1 around 100 ms after the stimulus, and for late components around 300-500 ms after the stimulus, particularly the P300.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques LUAUTE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No